CLINICAL TRIAL: NCT03480568
Title: A Phase III Trial to Evaluate the Efficacy and Safety of Biweekly Alirocumab in Patients on a Stable Dialysis Regimen: The Alidial Study
Brief Title: Alirocumab in Patients on a Stable Dialysis Regimen
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor Research Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018-038
Record Dates: First submitted 2018-03-01; First posted 2018-03-29 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Hemodialysis; Peritoneal Dialysis; Hypercholesterolemia; Atherosclerotic Disease
Keywords: Alirocumab
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: Open-label, nonrandomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- alirocumab (Experimental): Alirocumab 150 mg q 2 weeks for 12 weeks
  Interventions: Drug: Alirocumab 150 MG/ML [Praluent]

INTERVENTIONS:
Drug: Alirocumab 150 MG/ML [Praluent] — Cholesterol-lowering therapy

SUMMARY:
12-week study of the efficacy and safety of alirocumab in patients maintained stably on hemodialysis or peritoneal dialysis. Measures of cholesterol levels, drug levels, PCSK9 levels, routine chemistry and cell counts, and biomarkers will be obtained at baseline and at weeks 4, 8, 10 and 12 weeks. Safety events will be obtained throughout the study.

DETAILED DESCRIPTION:
Primary objective: The objective of this trial is to demonstrate the efficacy of alirocumab 150 mg every 2 weeks over 12 weeks on cholesterol levels.

Secondary objective: To assess the safety of treating chronic dialysis patients with alirocumab 150 mg subcutaneously every 2 weeks for 12 weeks.

Secondary objective: To demonstrate the efficacy of alirocumab 150 mg every 2 weeks over 12 weeks on biomarkers.

Exploratory objective: To assess alirocumab drug levels in subjects maintained on hemodialysis and peritoneal dialysis.

Methodology: Open-label, nonrandomized study

Number of patients Ten patients maintained on stable hemodialysis for a minimum of 3 months and ten patients maintained on stable peritoneal dialysis for a minimum of 3 months

Test product: alirocumab 150 mg

Mode of administration: administered subcutaneously

Dosing interval: every 2 weeks

Duration of treatment: 12 weeks

Primary endpoint: Levels of LDL-cholesterol at 12 weeks

Secondary endpoints: Levels of total cholesterol, triglycerides, apoprotein B, Cystatin-C, fibrinogen, hsCRP, IL-6, NGAL, NT-proBNP, soluble CD40 ligand, troponin T, VCAM

Safety criteria: Adverse events, Incidence and intensity of AE, including serious AE (SAE), Withdrawal from study medication due to AE, Clinical relevant new findings or worsening of existing conditions physical examination, Clinically relevant changes in laboratory measurements from baseline

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ages 18 to 80 years.
2. Written informed consent will be obtained before any study assessment is performed.
3. Diagnosis of end-stage renal disease, maintained on dialysis, without dialysis complications, for at least 3 months.
4. Patients may or may not have a diagnosis of atherosclerotic disease, such as a history of myocardial infarction (MI), cardiac percutaneous coronary intervention (PCI), coronary artery bypass (CABG) surgery, atherosclerotic transient ischemic attack (TIA) or cerebrovascular attack (CVA), or peripheral arterial disease (PAD).
5. A total of 20 patients will be enrolled, 10 patients on hemodialysis and 10 patients on peritoneal dialysis.

Exclusion Criteria:

1. LDL-cholesterol level of < 70 mg/dL.
2. Any contraindication to subcutaneous injections.
3. Patients on statin and/or ezetimibe therapy will have their cholesterol-lowering therapy continued as is without change during the time of the study.
4. History of any allergy or intolerance to the study drug or drugs of the same class.
5. A history of MI, PCI, CABG surgery, TIA, CVA, or PAD events within 3 months of enrollment.
6. History of malignant cancer within the past 3 years, excepting basal cell skin cancer or cervical cancer in situ.
7. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of the drug and for 2 weeks after the last injection of the drug. Highly effective methods of contraception include:

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
   3. Male sterilization (at least 6 months prior to enrollment). For female patients in the study, the vasectomized male partner should be the sole partner for that patient.
   4. Use of oral (estrogen and/or progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
   5. In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
   6. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before enrollment.
8. Pregnant or lactating women.
9. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or extraction of study drug, at investigator's discretion.
10. History or evidence of drug or alcohol abuse within the last 12 months.
11. Patients considered unsuitable for the study, including patients with psychiatric, behavioral or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in LDL cholesterol levels | Baseline, 4 ,8, 12 weeks
  Efficacy

SECONDARY OUTCOMES:
Change in HDL-cholesterol levels | Baseline, 12 weeks
  Efficacy
Change in apoprotein B levels | Baseline, 4, 8, 12 weeks
  Efficacy

OTHER OUTCOMES:
Change in PCSK9 levels | Baseline, 4, 8, 10, 12 weeks
  Efficacy
Change in alirocumab drug levels | Baseline, 4, 8, 10, 12 weeks
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Cara East, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Soltero CV Research, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Will provide data upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 6 weeks of request

REFERENCES:
- [Result] Collins AJ, Foley RN, Herzog C, Chavers BM, Gilbertson D, Ishani A, Kasiske BL, Liu J, Mau LW, McBean M, Murray A, St Peter W, Guo H, Li Q, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Dalleska F, Daniels F, Dunning S, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers PW, Agodoa L. Excerpts from the US Renal Data System 2009 Annual Data Report. Am J Kidney Dis. 2010 Jan;55(1 Suppl 1):S1-420, A6-7. doi: 10.1053/j.ajkd.2009.10.009. No abstract available. PMID 20082919
- [Result] van der Velde M, Matsushita K, Coresh J, Astor BC, Woodward M, Levey A, de Jong P, Gansevoort RT; Chronic Kidney Disease Prognosis Consortium; van der Velde M, Matsushita K, Coresh J, Astor BC, Woodward M, Levey AS, de Jong PE, Gansevoort RT, Levey A, El-Nahas M, Eckardt KU, Kasiske BL, Ninomiya T, Chalmers J, Macmahon S, Tonelli M, Hemmelgarn B, Sacks F, Curhan G, Collins AJ, Li S, Chen SC, Hawaii Cohort KP, Lee BJ, Ishani A, Neaton J, Svendsen K, Mann JF, Yusuf S, Teo KK, Gao P, Nelson RG, Knowler WC, Bilo HJ, Joosten H, Kleefstra N, Groenier KH, Auguste P, Veldhuis K, Wang Y, Camarata L, Thomas B, Manley T. Lower estimated glomerular filtration rate and higher albuminuria are associated with all-cause and cardiovascular mortality. A collaborative meta-analysis of high-risk population cohorts. Kidney Int. 2011 Jun;79(12):1341-52. doi: 10.1038/ki.2010.536. Epub 2011 Feb 9. PMID 21307840
- [Result] Rogacev KS, Pinsdorf T, Weingartner O, Gerhart MK, Welzel E, van Bentum K, Popp J, Menzner A, Fliser D, Lutjohann D, Heine GH. Cholesterol synthesis, cholesterol absorption, and mortality in hemodialysis patients. Clin J Am Soc Nephrol. 2012 Jun;7(6):943-8. doi: 10.2215/CJN.05170511. Epub 2012 Mar 29. PMID 22461539
- [Result] 6. KDIGO clinical practice guideline for lipid management in chronic kidney disease. Kidney Int Suppl. 2013;3:259-286.
- [Result] Chapter 2: Pharmacological cholesterol-lowering treatment in adults. Kidney Int Suppl (2011). 2013 Nov;3(3):271-279. doi: 10.1038/kisup.2013.34. No abstract available. PMID 25019001
- [Result] Kovesdy CP, Anderson JE, Kalantar-Zadeh K. Inverse association between lipid levels and mortality in men with chronic kidney disease who are not yet on dialysis: effects of case mix and the malnutrition-inflammation-cachexia syndrome. J Am Soc Nephrol. 2007 Jan;18(1):304-11. doi: 10.1681/ASN.2006060674. Epub 2006 Dec 13. PMID 17167114
- [Result] Shoji T. Serum lipids and prevention of atherosclerotic cardiovascular events in hemodialysis patients. Clin Exp Nephrol. 2014 Apr;18(2):257-60. doi: 10.1007/s10157-013-0871-z. Epub 2013 Sep 27. PMID 24072417
- [Result] Wanner C, Krane V, Marz W, Olschewski M, Mann JF, Ruf G, Ritz E; German Diabetes and Dialysis Study Investigators. Atorvastatin in patients with type 2 diabetes mellitus undergoing hemodialysis. N Engl J Med. 2005 Jul 21;353(3):238-48. doi: 10.1056/NEJMoa043545. PMID 16034009
- [Result] Marz W, Genser B, Drechsler C, Krane V, Grammer TB, Ritz E, Stojakovic T, Scharnagl H, Winkler K, Holme I, Holdaas H, Wanner C; German Diabetes and Dialysis Study Investigators. Atorvastatin and low-density lipoprotein cholesterol in type 2 diabetes mellitus patients on hemodialysis. Clin J Am Soc Nephrol. 2011 Jun;6(6):1316-25. doi: 10.2215/CJN.09121010. Epub 2011 Apr 14. PMID 21493741
- [Result] Krane V, Schmidt KR, Gutjahr-Lengsfeld LJ, Mann JF, Marz W, Swoboda F, Wanner C; 4D Study Investigators (the German Diabetes and Dialysis Study Investigators). Long-term effects following 4 years of randomized treatment with atorvastatin in patients with type 2 diabetes mellitus on hemodialysis. Kidney Int. 2016 Jun;89(6):1380-7. doi: 10.1016/j.kint.2015.12.033. Epub 2016 Feb 17. PMID 26924051
- [Result] Fellstrom BC, Jardine AG, Schmieder RE, Holdaas H, Bannister K, Beutler J, Chae DW, Chevaile A, Cobbe SM, Gronhagen-Riska C, De Lima JJ, Lins R, Mayer G, McMahon AW, Parving HH, Remuzzi G, Samuelsson O, Sonkodi S, Sci D, Suleymanlar G, Tsakiris D, Tesar V, Todorov V, Wiecek A, Wuthrich RP, Gottlow M, Johnsson E, Zannad F; AURORA Study Group. Rosuvastatin and cardiovascular events in patients undergoing hemodialysis. N Engl J Med. 2009 Apr 2;360(14):1395-407. doi: 10.1056/NEJMoa0810177. Epub 2009 Mar 30. PMID 19332456
- [Result] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Result] Everett BM, Smith RJ, Hiatt WR. Reducing LDL with PCSK9 Inhibitors--The Clinical Benefit of Lipid Drugs. N Engl J Med. 2015 Oct 22;373(17):1588-91. doi: 10.1056/NEJMp1508120. Epub 2015 Oct 7. No abstract available. PMID 26444323
- [Derived] East C, Bass K, Mehta A, Rahimighazikalayed G, Zurawski S, Bottiglieri T. Alirocumab and Lipid Levels, Inflammatory Biomarkers, Metabolomics, and Safety in Patients Receiving Maintenance Dialysis: The ALIrocumab in DIALysis Study (A Phase 3 Trial to Evaluate the Efficacy and Safety of Biweekly Alirocumab in Patients on a Stable Dialysis Regimen). Kidney Med. 2022 May 20;4(7):100483. doi: 10.1016/j.xkme.2022.100483. eCollection 2022 Jul. PMID 35801187
- See also: 1. Kidney disease statistics for the United States. Kidney.niddk.nih.gov. — https://www.niddk.nih.gov/health-information/health-statistics
- See also: 2. Statistics, The Kidney Project. Pharm.ucsf.edu/kidney/need/statistics. — https://pharm.ucsf.edu/kidney
- See also: 15. PCSK9 gene-genetics home reference. Ghr.nlm.nih.gov/gene/PCSK9. — https://ghr.nlm.nih.gov/gene/PCSK9